CLINICAL TRIAL: NCT02097589
Title: The Effect of Short-term Atorvastatin Treatment on Immune Responses to Pneumovax 23
Acronym: StatVax
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB201400208
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Controls
Keywords: Health Controls
MeSH Terms: interventions — Atorvastatin; 23-valent pneumococcal capsular polysaccharide vaccine; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pneumovax-Atorvastatin (Experimental): 10-person arm receiving treatment for 28 days: 40 mg atorvastatin, taken orally, once daily, for 28 days. Pneumovax 23 injected once, intramuscularly at Day 7.
  Interventions: Drug: Atorvastatin; Drug: Pneumovax 23
- Pneumovax-Placebo (Placebo Comparator): 10-person arm receiving treatment for 28 days: Placebo (lactose pill), taken orally, once daily for 28 days. Pneumovax 23 injected once, intramuscularly at Day 7.
  Interventions: Drug: Pneumovax 23; Other: Placebo (lactose pill)

INTERVENTIONS:
Drug: Atorvastatin — 10-person arm receiving treatment for 28 days: 40 mg atorvastatin, taken orally, once daily, for 28 days.
  Other Names: Lipitor
  Arms: Pneumovax-Atorvastatin
Drug: Pneumovax 23 — Pneumovax 23 injected once, intramuscularly at Day 7.
  Other Names: 23-valent pneumococcal polysaccharide vaccine
Other: Placebo (lactose pill) — 10-person arm receiving treatment for 28 days: Placebo (lactose pill), taken orally, once daily for 28 days.
  Arms: Pneumovax-Placebo

SUMMARY:
The purpose of this research study is to: Improve the effectiveness of vaccinations by identifying the effect of cholesterol medication, statins, on immune responses.

DETAILED DESCRIPTION:
Due to the anti-inflammatory action of statins, it was proposed that statin treatment would decrease the efficacy of vaccination. This response has yet to be explored following a primary vaccination such as pneumococcal pneumonia. In this study, healthy volunteers will be divided into 2 arms receiving treatment for 28 days: 40 mg atorvastatin or placebo.

Antibody titer for 23 serotypes, complete blood count (CBC), high-sensitivity c-reactive protein (hsCRP), erythrocyte sedimentation rate (ESR), lipids, cytokines (TNF-alpha, IFN-gamma, interleukins, etc.) and key membrane receptors (toll-like receptors, etc.) will be measured for baseline before statin or placebo treatment. On day 7 of treatment, pre-vaccination measures of the above parameters will be taken and an immune response will be induced in all groups using Pneumovax 23 at Day 7. On days 8, 14, 21, and 28 post-vaccination measures will be compared to baseline and between groups.

ELIGIBILITY:
Inclusion Criteria:

24 subjects are healthy volunteers between the ages of 21 and 40.

Exclusion Criteria:

1. Pregnant, planning to become pregnant, breastfeeding
2. Taking any of the following medications at time of study: antacids, antifungals, antioxidants, colestipol, cyclosporine, digoxin, erythromycin, fibric acid derivatives, niacin, oral contraceptives containing norethindrone or ethinyl estradiol, statins, steroids
3. Taking any immunosuppressive drugs including azathioprine, methotrexate, TNF inhibitors, cyclophosphamide, antimalarials, or sulfasalazine
4. Currently have or history of cardiovascular disease, diabetes, diphtheria, high blood pressure, high cholesterol, immunodeficiencies, kidney disease, liver disease, low blood pressure, muscular disease, seizure disorders, systemic lupus erythematosus or other systemic autoimmune disorders
5. Not immunized in childhood against streptococcus pneumoniae; received pneumovax vaccine within past year, or received 2 or more pneumovax boosters within the past 5 years
6. Latex allergy or previous allergic reaction or severe side effects from any vaccine
7. Heavy drinking (more than 15 drinks/week), illegal drug use within past six months, unwillingness to abstain from alcohol, unwillingness to abstain from tobacco products (dip, cigarettes, cigars, electronic cigarettes, etc.), illegal drugs, or grapefruit juice for duration of study
8. BMI over 30, abnormal values on lipid panel or liver function test
9. Failure to pass pre-study medical screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Determine the effect of atorvastatin treatment on pneumococcal antigen specific antibody production. | approximately 49 days
  The 24 subjects will be randomized into 2 groups of 12 individuals (6 per gender) and will be assigned to receive either atorvastatin treatment (40mg/day) or placebo (lactose pill) control.
  Subjects will be asked to fast after midnight prior to any morning blood draws. On day 1 of treatment, blood will be drawn for a baseline. Treatment with either atorvastatin or placebo will begin on day one and will continue until day 28. Subjects will be instructed to take the study medication once a day at the same time each day.
  On day seven of treatment, subjects will be immunized with Pneumovax 23, administered intramuscularly into the arm. Blood will be drawn at several time points following Pneumovax 23 administration. Measurements on blood will be made to determine the effect of statins on immune factor gene expression, serum protein levels, as well as at the cellular level.

SECONDARY OUTCOMES:
Determine the effect of atorvastatin treatment on immunogenic cytokine levels following pneumococcal vaccination. | approximately 49 days
  The 24 subjects will be randomized into 2 groups of 12 individuals (6 per gender) and will be assigned to receive either atorvastatin treatment (40mg/day) or placebo (lactose pill) control.
  Subjects will be asked to fast after midnight prior to any morning blood draws. On day 1 of treatment, blood will be drawn for a baseline. Treatment with either atorvastatin or placebo will begin on day one and will continue until day 28. Subjects will be instructed to take the study medication once a day at the same time each day.
  On day seven of treatment, subjects will be immunized with Pneumovax 23, administered intramuscularly into the arm. Blood will be drawn at several time points following Pneumovax 23 administration. Measurements on blood will be made to determine the effect of statins on immune factor gene expression, serum protein levels, as well as at the cellular level.

OTHER OUTCOMES:
Determine the effect of atorvastatin treatment on immune-regulatory gene expression. | Approximately 49 days
  The 24 subjects will be randomized into 2 groups of 12 individuals (6 per gender) and will be assigned to receive either atorvastatin treatment (40mg/day) or placebo (lactose pill) control.
  Subjects will be asked to fast after midnight prior to any morning blood draws. On day 1 of treatment, blood will be drawn for a baseline. Treatment with either atorvastatin or placebo will begin on day one and will continue until day 28. Subjects will be instructed to take the study medication once a day at the same time each day.
  On day seven of treatment, subjects will be immunized with Pneumovax 23, administered intramuscularly into the arm. Blood will be drawn at several time points following Pneumovax 23 administration. Measurements on blood will be made to determine the effect of statins on immune factor gene expression, serum protein levels, as well as at the cellular level.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Brantly, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Clinical Translational Research Building, Gainesville, Florida, United States

REFERENCES:
- [Derived] Wildes TJ, Grippin A, Fasanya H, Dyson KA, Brantly M. Effect of atorvastatin on humoral immune response to 23-valent pneumococcal polysaccharide vaccination in healthy volunteers: The StatVax randomized clinical trial. Vaccine. 2019 Feb 28;37(10):1313-1324. doi: 10.1016/j.vaccine.2019.01.023. Epub 2019 Jan 25. PMID 30686636